CLINICAL TRIAL: NCT06362174
Title: Capsule & Omics for pRedicting Exacerbation of Crohn's Disease (CORE-CD)
Brief Title: Capsule & Omics for pRedicting Exacerbation of Crohn's Disease
Acronym: CORE-CD
Status: Active, not recruiting | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Shomron BenHorin, Director of the Institute for Gastrointestinal Diseases (Gastrology), Sheba Medical Center
Other Study IDs: SHEBA-22-9902-SBH-CTIL
Record Dates: First submitted 2024-02-13; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies, fecal washes, stool samples and blood tests
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research group have previously evaluated the benefit of serial consecutive capsule endoscopy as monitoring tool for Crohn's disease in remission, demonstrating its superior accuracy for disclosing inflammation and for prediction of flares in comparison to other diagnostic modalities such as magnetic resonance enterography and inflammatory biomarkers. Subsequently, deep learning algorithms had developed to provide excellent accuracy for identification and grading of ulcers and intestinal strictures on capsule endoscopy still images. The investigators will advance this knowledge using a parallel two-parts approach.

DETAILED DESCRIPTION:
Part I - A retrospective study will use stored capsule and clinical datasets from 120 previously enrolled CD patients in remission, who underwent capsule based 24-months monitoring as part of two prior similar research projects (60 in each of the Israeli Inflammatory bowel disease Research Nucleus (IIRN), IIRN-I and IIRN-II-CURE- projects), aiming to predict and prevent flares based on capsule studies. The investigators will now utilize the accumulated visual data to develop AI-based complete film readouts and integrate the resultant visual omics data with previously derived microbiome and biomarker data, to serve as a discovery cohort for machine learning models predicting clinical exacerbation in patients in remission, which was witnessed in 27% of IIRN-I cohort within the 24m study.

Part II - A prospective observational study will enroll a new IIRN-III cohort of 60 (+6 attrition-considered) Crohn's Disease patients>16 years old in clinical remission. The investigators will deliberately use similar inclusion, monitoring design and outcome definitions as IIRN-I & II studies, to allow cross-cohort comparative validity. Procedures will include baseline colonoscopy, pan-enteric capsule and magnetic resonance enterography/Intestinal ultrasound, and thereafter serial capsule studies or every 6 months for 24 months. Newly acquired Omics will include baseline mucosal +colonic wash transcriptomics obtained during the baseline colonoscopy, serial dense stool microbiome and blood metabolomics, and a computerized frequency questionnaire, diet omics data. A densely sampled 24 months stool will be used to develop novel multi-omics tools predicting flares. The investigators will also use the datasets to explore the mechanisms and pathways involved in triggering remission transition into a clinical flare.

Follow- up can optionally extend to 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Age above 16
* Established Crohn's disease (CD) for at least 3 months
* Steroid free remission whether induced medically or surgically, for at least 3 months before inclusion
* CDAI<150
* Stable dose before enrollment:

  60 days for thiopurines, Methotrexate, Infliximab and Vedolizumab; 30 days for all other agents.

Exclusion Criteria:

* Corticosteroid use within the last 3 months
* Severe co-morbidities: liver, kidney, neurologic, metabolic or cardio-respiratory disorders not controlled at the time of enrollment
* Difficulty swallowing / history of aspirations or dysphagia
* Implanted metal objects precluding performance of MRI
* Cardiac pace-maker
* Known or suspected intestinal obstruction/stricture
* Pregnancy
* Alcohol / drug dependency
* Use of NSAIDs (including aspirin) for more than 3 continuous days, or during the 4 weeks preceding baseline visit.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Eligible patients will consist of adult CD patients >16YO in clinical remission, as determined by the validated Crohn's disease activity index (CDAI) of <150 and whose disease is known to involve the small bowel as either small bowel CD or ileo-colonic CD. Patients will have to be in steroid-free remission, whether induced medically or surgically, for at least 3 months before inclusion. Patients will be included regardless of the medication used for their treatment, but the dose of medication will be required to be stable before enrollment (60 days for thiopurines, Methotrexate, infliximab, vedolizumab, adalimumab and ustekinumab, 30 days for all other agents).
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Crohn's Disease Activity Index score (CDAI) | Score will be calculated every 3 months assessed up to 36 months. If score above 150 and a rise above 70 points from baseline patient will be withdrawn with clinical flare
  The rate of clinical relapse or disease complication by 24 months after inclusion defined as Crohn's Disease Activity Index above 150 and a rise above 70 points from pre flare value.
  Patients who experience CDAI score worsening without any other objective signs of disease inflammatory flare (i.e. without elevated C reactive protein (CRP) levels or elevated calprotectin levels or abnormal video capsule endoscopy (VCE) score) and without complication or change of CD medications - will be considered as primary outcome as per the original protocol definitions, but may be maintained on the study follow-up plan for the intended follow up period of 24 months or until 36 months.
Disease related complications | During hospitalization or after evaluation of tests results every 3 months, assessed up to 36 months
  onset of obstructive symptoms coupled with objective imaging and/or endoscopic evidence of new intestinal stricture, or occurrence of new penetrating complication.
disease related hospitalization | During hospitalization or after evaluation of tests results every 3 months, assessed up to 36 months.
  Disease related hospitalization in which patient was hospitalized due to disease related complications or flare.
Change of crohn's disease medications | Every 3 months, assessed up to 36 months.
  change of crohn's disease medications (type or dose)
opinion of the principle investigator (PI) or the treating physician | Every 3 months, assessed up to 36 months.
  Patients withdrawn due physician judgment of severity of mucosal lesions on video capsule endoscopy mandating change of therapy will be considered as non-responder (i.e. experienced a flare) for the purpose of the primary outcome.

SECONDARY OUTCOMES:
The rate of clinical flare accompanied by objective signs of mucosal inflammation. | through study completion, an average of 2 years.
  The later include Lewies score>350 + an increase of at least 225 Lewies score points from baseline on video capsule endoscopy study, OR a calprotectin above 250 with a at least 50% increase from baseline level, OR a C-Reactive Protein level more than X2 from upper limit of normal (ULN) for a patient with normal C-Reactive Protein at baseline.
The rate of inflammatory worsening with/without accompanying clinical symptoms | through study completion, an average of 2 years.
  defined as the occurrence of any of the aforementioned objective signs of mucosal inflammation

CONTACTS AND LOCATIONS:
Overall Officials: Shomron Ben- Horin, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel